CLINICAL TRIAL: NCT05484505
Title: Effectiveness of Preloaded Combination Nicotine Replacement Therapy on Smoking Cessation of Adult Population in Kazakhstan- A Randomized Controlled Trial
Brief Title: Preloaded Combination Nicotine Replacement Therapy on Smoking Cessation of Adult Population in Kazakhstan
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nazarbayev University (Other)
Collaborators: Astana Medical University (Other)
Responsible Party: Principal Investigator, Chethan Purushothama, Assistant Professor, Nazarbayev University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11022021CRP1514
Record Dates: First submitted 2022-07-22; First posted 2022-08-02 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Smoking Cessation; Smoking, Cigarette; Smoking Behaviors
Keywords: Tobacco; Smoking; Nicotine Patches; Nicotine Gums; Nicotine Replacement Therapy; Preloading
MeSH Terms: conditions — Smoking Cessation; Cigarette Smoking; Smoking | interventions — Tobacco Use Cessation Devices; Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine replacement therapy (NRT) Preloading (Experimental): 1. Brief Advice (5 A's & 5 R's)- 0-day, Month- 1, 3, 6, 9, 12
  2. a. Nicotine Replacement Therapy for > 20 cigarettes per day
  Nicotine Patch: Preloading for 4 weeks + 12 weeks post quit date,21 mg: 4 weeks before and after quit date,14 mg: Next 4 weeks,7 mg: Last 4 weeks Nicotine chewing gums 4 mg for 12 weeks post quit date (12/day on week 1(Tapering dose weekly)1/day on week 12
  2.b. Nicotine Replacement Therapy for < 20 cigarettes per day Nicotine Patch: Preloading for 4 weeks + 12 weeks post quit date 21 mg: 4 weeks before and after quit date 14 mg: Next 4 weeks 7 mg: Last 4 weeks
  Nicotine chewing gums 2 mg for 12 weeks post quit date (12/day on week
  1(Tapering dose)1/day on week 12
  Interventions: Drug: Nicotine patch, Nicotine gums; Behavioral: Brief Advice (5 A's & 5 R's); Drug: Nicotine Patch: Preloading for 4 weeks
- Nicotine replacement therapy (NRT) (Active Comparator): 1. Brief Advice (5 A's & 5 R's)- 0-day, Month- 1, 3, 6, 9, 12
  2. a. Nicotine Replacement Therapy for > 20 cigarettes per day
  Nicotine Patch: 12 weeks post quit date 21 mg: 4 weeks after quit date 14 mg: Next 4 weeks 7 mg: Last 4 weeks
  Nicotine chewing gums 4 mg for 12 weeks post quit date (12/day on week 1(Tapering dose weekly)1/day on week 12
  2.b. Nicotine Replacement Therapy for < 20 cigarettes per day
  Nicotine Patch: 12 weeks post quit date 21 mg: 4 weeks after quit date 14 mg: Next 4 weeks 7 mg: Last 4 weeks
  Nicotine chewing gums 2 mg for 12 weeks post quit date (12/day on week 1(Tapering dose)1/day on week 12
  Interventions: Drug: Nicotine patch, Nicotine gums; Behavioral: Brief Advice (5 A's & 5 R's)

INTERVENTIONS:
Drug: Nicotine patch, Nicotine gums — Nicotine patch 21mg, 12 weeks post quit date and nicotine chewing gums 4mg for 12 weeks post quit date
  * 14 mg: Next 4 weeks
  * 7 mg: Last 4 weeks
  Other Names: Nicotex
Behavioral: Brief Advice (5 A's & 5 R's) — Brief Advice (5 A's & 5 R's) at Day 0, 1 month, 3,6,9 & 12 months
Drug: Nicotine Patch: Preloading for 4 weeks — Nicotine Patch: Preloading for 4 weeks - 21 mg: 4 weeks before quit date
  Arms: Nicotine replacement therapy (NRT) Preloading

SUMMARY:
Randomized, controlled, two-armed, single-blinded, superiority trial with 1:1 allocation ratio Nicotine Replacement Therapy(NRT)

DETAILED DESCRIPTION:
The primary objective is to determine the effectiveness of preloaded combination nicotine replacement therapy (NRT) on smoking cessation of tobacco smokers. The secondary objectives are to determine the predictors of smoking cessation among the study participant's, to determine the change in health-related quality of life due to smoking cessation & to determine the perception of treatment adherence among the study participants.

ELIGIBILITY:
Inclusion Criteria:

* all current smokers aged 18 years and above with a motivation to quit

Exclusion Criteria:

* smokeless tobacco users, smoking frequency of fewer than 10 cigarettes per day, pregnant women, lactating women, patients with a recent history of myocardial infarction of fewer than 3 months, and electronic cigarette users

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Self reported smoking during intervention period : Yes/No | Assessed at 12 months from the starting point of intervention.
  Self-reported smoking anytime during the intervention or follow-up period
Salivary cotinine test results: Positive or Negative | Salivary cotinine test results before intervention, after the intervention and after follow ups
  Salivary cotinine test results before, during and after the intervention

SECONDARY OUTCOMES:
Self reported number of quit attempts of tobacco | Assessed at 3, 6 & 12 months from the starting point of intervention.
  Number of quit attempts of tobacco since enrolment
Self reported number of smoked cigarettes/bidis per day | Assessed at 12 months from the starting point of intervention.
  Number of smoked cigarettes/bidis per day since enrolment
Adherence to intervention in days: Self reported | Assessed at 12 months from the starting point of intervention.
  Self reported duration of use of the intervention in days

OTHER OUTCOMES:
Pattern of smoking | Assessed at 12 months from the starting point of intervention.
  The change in smoking frequency from the baseline information (It can be excess use, reduced use or relapse)

CONTACTS AND LOCATIONS:
Locations (2):
- Kazakhstan (2):
  - National Research Cardiac Surgery Center, Astana, Kazakhstan, Astana
  - Nazarbayev University School of Medicine, Astana

IPD SHARING:
Plan to Share IPD: Yes
The data of the current study will available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from the corresponding author on reasonable request.
Access Criteria: Data will be available from the corresponding author on reasonable request via e-mail

REFERENCES:
- [Result] Hays JT, Croghan IT, Baker CL, Cappelleri JC, Bushmakin AG. Changes in health-related quality of life with smoking cessation treatment. Eur J Public Health. 2012 Apr;22(2):224-9. doi: 10.1093/eurpub/ckq137. Epub 2010 Sep 30. PMID 20884658
- [Result] Wang Q, Mati K. Intention to Quit among Smokers in Kazakhstan: Data from 2014 Global Adult Tobacco Survey. J Epidemiol Glob Health. 2019 Mar;9(1):23-28. doi: 10.2991/jegh.k.190212.002. PMID 30932386
- [Result] Levy DT, Levy J, Mauer-Stender K. Potential impact of strong tobacco-control policies in 11 newly independent states. Cent Eur J Public Health. 2019 Jun;27(2):115-126. doi: 10.21101/cejph.a5506. PMID 31241286
- [Result] Giulietti F, Filipponi A, Rosettani G, Giordano P, Iacoacci C, Spannella F, Sarzani R. Pharmacological Approach to Smoking Cessation: An Updated Review for Daily Clinical Practice. High Blood Press Cardiovasc Prev. 2020 Oct;27(5):349-362. doi: 10.1007/s40292-020-00396-9. Epub 2020 Jun 23. PMID 32578165
- [Result] Llimargas M, Lawrence PA. Seven Wnt homologues in Drosophila: a case study of the developing tracheae. Proc Natl Acad Sci U S A. 2001 Dec 4;98(25):14487-92. doi: 10.1073/pnas.251304398. Epub 2001 Nov 20. PMID 11717401
- [Result] Prochaska JJ. Nicotine Replacement Therapy as a Maintenance Treatment. JAMA. 2015 Aug 18;314(7):718-9. doi: 10.1001/jama.2015.7460. PMID 26284723
- [Result] Chai W, Zou G, Shi J, Chen W, Gong X, Wei X, Ling L. Evaluation of the effectiveness of a WHO-5A model based comprehensive tobacco control program among migrant workers in Guangdong, China: a pilot study. BMC Public Health. 2018 Feb 27;18(1):296. doi: 10.1186/s12889-018-5182-6. PMID 29486753
- [Result] Dhavan P, Bassi S, Stigler MH, Arora M, Gupta VK, Perry CL, Ramakrishnan L, Reddy KS. Using salivary cotinine to validate self-reports of tobacco use by Indian youth living in low-income neighborhoods. Asian Pac J Cancer Prev. 2011;12(10):2551-4. PMID 22320954
- [Result] Rose JE, Behm FM, Westman EC. Nicotine-mecamylamine treatment for smoking cessation: the role of pre-cessation therapy. Exp Clin Psychopharmacol. 1998 Aug;6(3):331-43. doi: 10.1037//1064-1297.6.3.331. PMID 9725117
- [Result] Hymowitz N, Cummings KM, Hyland A, Lynn WR, Pechacek TF, Hartwell TD. Predictors of smoking cessation in a cohort of adult smokers followed for five years. Tob Control. 1997;6 Suppl 2(Suppl 2):S57-62. doi: 10.1136/tc.6.suppl_2.s57. PMID 9583654
- [Derived] Purushothama C, Crape BL, Stolyarov V, Jaxybayeva A, la Fleur P, Olickal JJ. Preloaded combination nicotine replacement therapy for smoking cessation in Kazakhstan: A randomized controlled trial study protocol. PLoS One. 2023 Nov 27;18(11):e0292490. doi: 10.1371/journal.pone.0292490. eCollection 2023. PMID 38011129
- See also: Carbon monoxide breath analyzers and its role in tobacco cessation: A narrative review of literature. — https://www.jioh.org/text.asp?2018/10/2/71/230862